CLINICAL TRIAL: NCT03672669
Title: Comparison of the Effect of Advanced Platelet-rich Fibrin and Leukocyte- and Platelet-rich Fibrin on Outcomes After Removal of Impacted Mandibular Third Molar: A Randomised Split-mouth Study
Brief Title: Comparison of the Effect of A-PRF and L-PRF on Outcomes After Removal of Impacted Mandibular Third Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Mehmet Gagari Caymaz, Research Assistant, Near East University, Turkey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Near East University
Record Dates: First submitted 2018-09-11; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Pain, Postoperative; Trismus; Swelling
Keywords: Leukocyte- and platelet rich fibrin; Advanced platelet rich fibrin; Impacted mandibular third molar surgery
MeSH Terms: conditions — Pain, Postoperative; Trismus | interventions — Leukocyte Count

STUDY DESIGN:
Intervention Model Description: patients with bilateral impacted mandibular third molar which surgically operated at different times
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Platelet Rich Fibrin (A-PRF) (Active Comparator): A-PRF was applied into the tooth socket after mandibular third molar surgery.
  Interventions: Genetic: Advanced Platelet Rich Fibrin (A-PRF)
- Leukocyte- and platelet-rich fibrin (L-PRF) (Active Comparator): L-PRF was applied into the tooth socket after mandibular third molar surgery.
  Interventions: Genetic: Leukocyte- and platelet-rich fibrin (L-PRF)

INTERVENTIONS:
Genetic: Advanced Platelet Rich Fibrin (A-PRF) — blood samples collected in 10 ml of vacuumed plain glass tubes were centrifuged for 14 minutes at 1500 rpm without anticoagulant agents in order to obtain A-PRF
  Arms: Advanced Platelet Rich Fibrin (A-PRF)
Genetic: Leukocyte- and platelet-rich fibrin (L-PRF) — blood samples collected in 10 ml of glass coated plastic tubes were centrifuged without anticoagulant agents for 10 minutes in order to obtain L-PRF
  Arms: Leukocyte- and platelet-rich fibrin (L-PRF)

SUMMARY:
In this study, it was aimed to investigating and comparing the postoperative effects of leukocyte- and platelet-rich fibrin (L-PRF) and advanced platelet-rich fibrin (A-PRF) in terms of pain, swelling on the cheek, and trismus after mandibular third molar surgery. The study included a total of 27 patients with bilateral impacted mandibular third molar which surgically operated at different times. Patients were evaluated in two randomly separated groups. For the first group; A-PRF and for the second group; L-PRF was applied into the tooth socket. The outcomes variables were; pain, swelling, the number of analgesics taken, and trismus. These variables were also assessed on the basis of; 1st, 2nd, 3rd and 7th days following the operation.

ELIGIBILITY:
Inclusion Criteria:

* age≥18
* the presence of bilaterally symmetrically impacted mandibular third molar, which requires an extraction for prophylactic reasons
* absence of systemic diseases
* absence of chronic opioid taken;
* not being pregnant
* not smoking and no alcohol usage
* the absence of allergy to penicillin or any other drugs used during standardized postoperative therapy.

Exclusion Criteria:

* tooth needed to be sectioning during the operation
* operation time exceeding 30 minutes
* the cases with severe periodontal disease or acute pericoronitis,
* the cases using antibiotics for an existing infection
* the cases not capable of following postoperative instructions

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
Pain Scores Evaluted | 1st day after the operation.
  For the postoperative period, the pain scores change was evaluated with the help of the visual analog scale (VAS) ranging from 0 (no pain) to 10 (most severe pain).
Pain Scores Evaluted | 2nd day after the operation.
  For the postoperative period, the pain scores change was evaluated with the help of the visual analog scale (VAS) ranging from 0 (no pain) to 10 (most severe pain).
Pain Scores Evaluted | 3rd day after the operation.
  For the postoperative period, the pain scores change was evaluated with the help of the visual analog scale (VAS) ranging from 0 (no pain) to 10 (most severe pain).
Pain Scores Evaluted | 7th day after the operation.
  For the postoperative period, the pain scores change was evaluated with the help of the visual analog scale (VAS) ranging from 0 (no pain) to 10 (most severe pain).

SECONDARY OUTCOMES:
Number of Analgesics Taken by the Patients | Each patient was evaluated on the 1st, 2nd, 3rd, and 7th days after the operation.
Trismus | Each patient was evaluated in order to obtain measurements on the 1st, 2nd, 3rd, and 7th days after the operation.
  Trismus was assessed by measuring the distance between the mesioincisal corner of the maxillary and mandibular right incisors while mouth was fully opened
Swelling on the cheek | Each patient was evaluated in order to obtain measurements on the 1st, 2nd, 3rd, and 7th days after the operation.
  In order to record swelling, a modification of the tape measurement method

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet G Caymaz, DDS, Principal Investigator — Near East University
Locations (1):
- Near East University, Mersin, Turkey (Türkiye)